CLINICAL TRIAL: NCT01114867
Title: Prospective Cross-sectional Study of Fetal Penis and Corpus Cavernosum Length
Brief Title: Fetal Penile Length and Corpus Cavernosum Length - Normal Measurement Via Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yoseph Hartoov / Dr, Sorasky Medical Center
Other Study IDs: TASMC-10-YH-0128-CTIL
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2010-04

CONDITIONS: Fetal Penis Length
Keywords: ultrasound; penis length; corpus cavernosum; length of fetal penis and fetal corpus cavernosum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Measurement of fetal penis length by ultrasound may be inaccurate when measured from the scrotum to the penile tip. we will provide normal values of penile length measured from the penile tip to the abdominal wall and measuring the corpus cavernosum length.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 14th through 34th week gestation,
* routine ultrasound not preformed for anomalies at the genitourinary system,
* estimated fetal weight corresponds to gestational age.

Exclusion Criteria:

* women who's fetuses are suspected to be with fetal growth retardation,
* women who's fetuses are suspected to be with genitourinary anomaly.

Ages: 14 Weeks to 34 Weeks | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fetuses of healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Hartoov, Dr, Principal Investigator — Tel-Aviv, Soraski Medical Center
Locations (1):
- Ultrasound Unit in OBGYN, Soraski Medical Center, Tel Aviv, Israel